CLINICAL TRIAL: NCT01358318
Title: Effect of Addition of Soy Protein and Soy Fiber to a Snack Bar on Satiety and Food Intake
Brief Title: Effects of Soy Protein/Soy Fiber on Measures of Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solae, LLC (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GIL1103
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Lack of Satiety
Keywords: obesity; satiety; soy protein; soy fiber; control appetite; reduce food intake
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Control (Placebo Comparator)
  Interventions: Other: Satiety
- Soy Protein (Experimental)
  Interventions: Other: Satiety
- Soy Fiber (Experimental)
  Interventions: Other: Satiety
- Soy Protein and Soy Fiber (Experimental)
  Interventions: Other: Satiety

INTERVENTIONS:
Other: Satiety — Single consumption of snack bars to determine satiety and food intake at next meal.

SUMMARY:
The purpose of this study is to determine whether ingestion of a bar containing either added soy protein or soy fiber or both, increases subjective and objective measures of satiety compared to a control bar.

DETAILED DESCRIPTION:
The study will use a randomized, double blind crossover design in which subjects act as their own control. Satiation will be assessed using a Motivation to Eat Questionnaire. Height and weight will be measured at the screening visit and weight alone at each subsequent visit. Prior to consumption of the test meal (breakfast) and at 15, 30, 60, 90, 120 and 150 min thereafter, subjects will complete a VAS Motivation to Eat Questionnaire. After subjects complete the first VAS motivation questionnaire, they will be given the test meal and instructed to eat this over a 15 minute period and fill out a palatability questionnaire. Two hours after the start of the test meal they will be taken to a private feeding room, where an ad libitum pizza lunch will be served with mineral water. Participants will be instructed to eat and drink as much as they desire until they are comfortably full. Subjects will be asked to fill out a final VAS Motivation to eat questionnaire 30 min after the start of the pizza meal.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 30 kg/m2
* Age between 20-60y
* Unrestrained eater (score<15)
* Regularly consume 3 meals per day
* Moderate exercise (eg running , aerobics classes, other sports activities) of no more than 7 hours per week

Exclusion Criteria:

* use of drugs that influence carbohydrate or lipid metabolism (eg betablockers,hypoglycemic agents, antibiotics taken less than 6 weeks before study entry, glucocorticoids, anti-diarrheal medication, weight loss medication etc), and anti-diabetic medication
* presence of any significant disease (eg gastrointestinal diseases, diabetes, a CVD event less than 12 weeks from study entry, current hepatic disease etc)
* use of special dietary treatments or supplement within 4 weeks of study
* restrained eater (score>15)
* weight change (±10% of body weight) within the previous 6 weeks
* alcohol intake >2 drinks/day
* food allergies of any kind
* swallowing difficulties,
* exercising more than 7 hours per week

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Satiety | at each visit (4 visits total)
  visual analog scales for satiety

SECONDARY OUTCOMES:
Ad Libitum Energy Intake | at each visit (4 visits total)
  Pizza lunch amount consumed will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, PhD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada